CLINICAL TRIAL: NCT05459844
Title: A Study Comparing Treatment With Lutetium[177Lu] Oxodotreotide Injection to Octreotide LAR in Patients With Inoperable, Progressive, Well Differentiated, Somatostatin Receptor Positive Gastroenteropancreatic Neuroendocrine Tumours
Brief Title: A Study Comparing Treatment With Lutetium[177Lu] Oxodotreotide Injection to Octreotide LAR in Patients With GEP-NETs
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XT-XTR008-3-01
Record Dates: First submitted 2022-07-05; First posted 2022-07-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine tumour; 177Lu-Dota0-Tyr3-octreotate
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lutetium[177Lu] Oxodotreotide Injection (Experimental): Treatment consisted of a cumulative administered radioactivity of 29.6 Giga Becquerel (GBq) (800 mCi) Lutetium[177Lu] Oxodotreotide Injection: Four administrations of 7.4 GBq (200 mCi).
  Concomitant amino acids were given with each administration for kidney protection.
  Lutetium[177Lu] Oxodotreotide Injection was administered at 8 +/- 1-week intervals, which could be extended up to 16 weeks to accommodate resolving acute toxicity.
  In case participants experienced clinical symptoms (i.e. diarrhoea and flushing) associated with their carcinoid tumours, Octreotide s.c. rescue injections were allowed.
  Interventions: Drug: Lutetium[177Lu] Oxodotreotide Injection
- Octreotide LAR (Active Comparator): 60 mg Octreotide LAR treatment every 4 weeks (i.m. injections) until the end of the study, unless the participant progressed or died.
  In case participants experienced clinical symptoms (i.e. diarrhoea and flushing) associated with their carcinoid tumours, s.c. Octreotide rescue injections were allowed.
  Interventions: Drug: Octreotide LAR

INTERVENTIONS:
Drug: Lutetium[177Lu] Oxodotreotide Injection — Four administrations of 7.4 GBq (200 mCi) Lutetium[177Lu] Oxodotreotide Injection administered at 8 +/- 1-week intervals, which could be extended up to 16 weeks to accommodate resolving acute toxicity.
  Other Names: 177Lu-DOTA0-Tyr3-Octreotate
  Arms: Lutetium[177Lu] Oxodotreotide Injection
Drug: Octreotide LAR — 60 mg Octreotide LAR treatment was given to the participants every 4 weeks (i.m. injections) until the end of the study, unless the participant progressed or died.
  Other Names: SANDOSTATIN LAR, Octreotide
  Arms: Octreotide LAR

SUMMARY:
This was a multicenter, stratified, open, randomized, comparator-controlled, parallel-group phase III study comparing treatment with Lutetium[177Lu] Oxodotreotide Injection to high dose (60 mg) Octreotide LAR in patients with unresectable or metastatic, progressive, well differentiated (G1 and G2), somatostatin receptor positive gastroenteropancreatic neuroendocrine tumours.

DETAILED DESCRIPTION:
After the screening period, participants who signed the ICF and were eligible for the study in accordance with the entry criteria were randomly assigned to treatment either Lutetium[177Lu] Oxodotreotide Injection or Octreotide LAR. Participant randomization was performed according to a centralized permuted block randomization scheme with a balanced ratio (1:1) between the 2 treatment groups, stratified by primary site of tumor (pancreatic or non-pancreatic), NET pathological grading (G1 or G2) and by the length of time that a participant was on a constant dose of Octreotide (=< 6 versus > 6 months). Objective tumor assessment in both groups was performed every 12+/-1 weeks from the randomization date according to RECIST Criteria until progression was centrally confirmed: any participants with progressive disease ceased the treatment/assessment period and proceeded to the long-term follow-up period for evaluation of survival and long-term safety.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Aged 18 years or older.
3. Histopathologically confirmed low and moderate grade (G1 or G2) unresectable locally advanced or metastatic GEP-NET (based on the fifth edition of the WHO classification and grading criteria for neuroendocrine tumors of the digestive system in 2019, to be centrally confirmed).
4. Previously received fixed-dose Octreotide LAR (20-30 mg/3-4 weeks) for at least 12 weeks of continuous treatment with disease progression.
5. Presence of disease progression prior to randomization (time point of disease progression limited to 1 year prior to randomization and no other antitumor therapy received after progression).
6. Presence of at least 1 measurable site of disease (based on RECIST 1.1).
7. All target lesions (based on RECIST 1.1) at baseline must be confirmed as somatostatin receptor positive by 68Ga-Dotatate PET/CT .
8. ECOG score of 0 or 1.
9. Subjects of childbearing potential voluntarily use an effective method of contraception, such as condoms, oral or injectable contraceptives, IUDs, etc., during treatment and within 4 months (men) or 7 months (women) of the last use of the trial drug.

Exclusion Criteria:

1. Serum creatinine >150 μmol/L (1.7 mg/dL) or creatinine clearance <50 ml/min (Cockcroft Gault formula).
2. Hemoglobin <80g/L, or white blood cell count <2.0×10^9/L, or platelets <75×10^9/L.
3. Serum total bilirubin > 3 × upper limit of normal (ULN).
4. Serum albumin <30g/L.
5. alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5×ULN.
6. international normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 x ULN.
7. Positive human immunodeficiency virus (HIV) antibody.
8. Positive for hepatitis B virus (HBV) surface antigen (HBsAg) and positive for HBV DNA (≥1×10^4 copies/ml or judged positive by research center criteria), or positive for hepatitis C virus (HCV) antibodies.
9. Pregnant or lactating females.
10. Received peptide receptor radionuclide therapy(PRRT) prior to randomization.
11. Received Octreotide LAR at a dose strength >30 mg/3-4 weeks (increasing dose or frequency) within 12 weeks prior to randomization.
12. Any patient receiving treatment with short-acting Octreotide, which cannot be interrupted for 24 h before and 24 h after the administration of Lutetium[177Lu] Oxodotreotide Injection, or any patient receiving treatment with Octreotide LAR, which cannot be interrupted for at least 6 weeks before the administration of Lutetium[177Lu] Oxodotreotide Injection.
13. Received systemic antitumor therapy such as targeted therapy, immunotherapy, antitumor herbal therapy, chemotherapy within 4 weeks prior to randomization.
14. Participated in other drug clinical trials within 4 weeks prior to randomization and received treatment with the corresponding trial drug.
15. Received the following treatments within 12 weeks prior to randomization, including but not limited to surgery (except biopsy), radical radiotherapy, hepatic artery interventional embolization, cryoablation of liver metastases, or radiofrequency ablation.
16. Received external beam radiation therapy for bone metastases within 2 weeks prior to randomization
17. Toxicity of prior antitumor therapy has not returned to ≤ grade 1 levels (except for alopecia)
18. Known brain metastases, unless these metastases have been treated and stabilized for at least 24 weeks, prior to enrollment in the study.
19. Uncontrolled congestive heart failure, including baseline left ventricular ejection fraction (LVEF) <50%.
20. uncontrolled diabetes mellitus, including baseline fasting glucose > 2 x ULN.
21. Any clinically significant active infection.
22. Known other malignancies (except for those without recurrence within 5 years after adequate treatment)
23. Known hypersensitivity to Lutetium[177Lu] Oxodotreotide Injection or oxytetracycline acetate microsphere components and their excipients.
24. Known to be unsuitable for enhanced CT or MRI contrast imaging due to allergic reaction or renal insufficiency.
25. Any other disease, mental status or surgical condition that is uncontrolled, may interfere with study completion (including poor compliance) or is inappropriate for the use of the investigational drug.
26. Other treatment options (e.g., chemotherapy, targeted therapy) that, in the opinion of the investigator, are more appropriate for the patient than the treatment provided in the study based on the patient's disease characteristics, i.e., the investigational drug is not the best therapeutic agent for clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by BIRC | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  Progression Free Survival (PFS) was defined as the time from randomization to documented centrally assessed disease progression, as evaluated by the Blinded Independent Review Committee (BIRC), or death due to any cause. If a participant had no centrally assessed progression and had not died at the time of the primary endpoint analysis, the participant was regarded as censored in the context of a time to event analysis at the date of last evaluable tumor assessment. Disease progression was determined by objective tumor response status using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) assessed by investigator | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  Progression Free Survival (PFS) was defined as the time from randomization to documented investigator-assessed disease progression, or death due to any cause. If a participant had no investigator-assessed progression and had not died at the time of the primary endpoint analysis, the participant was regarded as censored in the context of a time to event analysis at the date of last evaluable tumor assessment. Disease progression was determined by objective tumor response status using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1).
Objective Response Rate (ORR) assessed by investigator | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  Objective Response Rate (ORR) was calculated as the proportion of patients with tumour size reduction (sum of partial responses (PR) and complete responses (CR)) and assessed by investigator according to RECIST 1.1.
Objective Response Rate (ORR) assessed by BIRC | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  Objective Response Rate (ORR) was calculated as the proportion of patients with tumour size reduction (sum of partial responses (PR) and complete responses (CR)) assessed by BIRC according to RECIST 1.1.
Duration of Response (DoR) assessed by investigator | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  The Duration of Response (DoR) was defined as the time from initially meeting the criteria for response (CR or PR) until the time of progression and assessed by investigator according to RECIST 1.1.
Duration of Response (DoR) assessed by BIRC | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  The Duration of Response (DoR) was defined as the time from initially meeting the criteria for response (CR or PR) until the time of progression assessed by BIRC according to RECIST v1.1.
Time to Tumour Progression (TTP) assessed by investigator | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  Time to Tumour Progression (TTP) was defined as the time from randomization to progression assessed by investigator. It included patients who dropped out due to toxicity, but omitted patients who died without measured progression (censored to last follow-up date or death date).
Time to Tumour Progression (TTP) assessed by BIRC | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  Time to Tumour Progression (TTP) was defined as the time from randomization to progression assessed by BIRC. It included patients who dropped out due to toxicity, but omitted patients who died without measured progression (censored to last follow-up date or death date).
Disease Control Rate (DCR) assessed by investigator | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  DCR is defined as the incidence of complete response, partial response and stable disease assessed by investigator according to RECIST v1.1.
Disease Control Rate (DCR) assessed by BIRC | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  DCR is defined as the incidence of complete response, partial response and stable disease assessed by BIRC according to RECIST v1.1.
20-month Progression-Free Survival rate assessed by BIRC | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  20-month Progression-Free Survival rate was defined as the proportion of patients whose time from randomization to disease progression by BIRC according to RECIST v1.1 or death exceeds 20 months.
20-month Progression-Free Survival rate assessed by investigator | From date of randomization until date of progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  20-month Progression-Free Survival rate was defined as the proportion of patients whose time from randomization to disease progression by investigator according to RECIST v1.1 or death exceeds 20 months.
Overall Survival (OS) | From date of randomization until date of death from any cause up to final safety cut-off date reached，assessed up to approximately 60 months
  Overall Survival (OS) was defined as the time from the date of randomization to the date of death due to any cause or the date of last contact (censored observation) prior to the date of the data cut-off, and during the entire study period (i.e. the treatment period plus follow-up).
Change From Baseline in the EORTC QLQ-C30 Questionnaire | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  The Quality of Life Questionnaire C30 (QLQ-C30) was developed by the European Organization for Research and Treatment of Cancer (EORTC) to assess quality of life in cancer patients. It includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality-of-life and financial impact. Subjects respond on a four-point scale from "not at all" to "very much" for most items. Raw scores are linearly transformed so each score ranged a 0-100, where higher scores indicate worse symptoms (e.g., more severe/worsened) and lower scores indicate less symptoms (e.g., less severe/improvement).
Change From Baseline in the EORTC Quality of Life Questionnaire - Neuroendocrine Carcinoid Module (EORTC QLQ-GINET21) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first until Primary Analysis cutoff date reached，assessed up to approximately 34 months
  The Quality of Life GI Neuroendocrine Tumor survey (QLQ GINET21) contains a total of 21 items: four single-item assessments relating to muscle and/or bone pain (MBP), body image (BI), information (INF) and sexual functioning (SX), together with 17 items organized into five proposed scales: endocrine symptoms (ED; three items), GI symptoms (GI; five items), treatment-related symptoms (TR; three items), social functioning (SF) and disease-related worries (DRW; three items). The response format of the questionnaire is a four-point Likert scale. Responses are linearly transformed to a 0-100 scale using EORTC guidelines, with higher scores reflecting more severe symptoms.
Number of Participants With Adverse Events | From informed consent signature through study completion reached at final safety cutoff date，assessed up to approximately 60 months
  The distribution of adverse events was done via the analysis of frequencies for Adverse Event (AEs), Serious Adverse Event (SAEs) and Deaths, through the monitoring of relevant clinical and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Principal Investigator — Chinese PLA General Hospital
Locations (23):
- China (23):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Afilliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of AFMU, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu F, Li P, Xu J, Zhang J, Xu X, Chen Z, Qiao Y, Liang Y, Chen J, Song S. Radiation exposure and protection advice after [177Lu]Lu-DOTA-TATE therapy in China. EJNMMI Res. 2024 Nov 28;14(1):119. doi: 10.1186/s13550-024-01185-4. PMID 39607652